CLINICAL TRIAL: NCT04425551
Title: Prospective Study of the Effect of Micropulse Laser on Dry Eye Disease Due to Meibomian Gland Dysfunction
Brief Title: Effect of Micropulse Laser on Dry Eye Disease Due to Meibomian Gland Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Naval Hospital, Athens (Other)
Collaborators: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Nikolaos Kappos, Ophthalmologist Surgeon, Clinical Investigator, Naval Hospital, Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 6/19
Record Dates: First submitted 2020-06-04; First posted 2020-06-11 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Dry Eye; Dry Eye Syndromes; Meibomian Gland Dysfunction
Keywords: dry eye; meibomian gland dysfunction; subthreshold laser; telangiectasia; eyelid margin vascularity
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction; Telangiectasis | interventions — Lasers

STUDY DESIGN:
Intervention Model Description: Please note that there was one group of participants, but two groups of eyes (treated/untreated). Thus, PARALLEL was selected, referring to eyes, not participants
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser Group (Active Comparator): The treatment involved laser photocoagulation of the telangiectatic vessels of the lower eyelid margin with a slit lamp-based 532 nm optically pumped dual- diode solid-state subthreshold (SP-Mode) laser system (LightLas TruScan Pro 532 nm, LightMed Corporation, San Clemente, CA, USA). The laser settings were selected to induce vascular photocoagulation without visible tissue blanching or epithelial disruption. The subthreshold treatment parameters were set at 50 μm spot size and duration of 200 ms with duty cycle of 20%. Laser power was titrated in mono-spot micropulse mode starting at 500 mW and increased in 100 mW steps, until focal blanching without epithelial whitening, maximum 1500 mW. The treatment endpoint was defined as immediate focal blanching (disappearance of the red reflex) of the target telangiectatic vessel, assessed under a high-magnification slit-lamp view, with the effect confined to the targeted vessel and no visible impact on adjacent tissue.
  Interventions: Procedure: laser light
- Control Group (Placebo Comparator): Sham treatment replicated all procedural steps (eyelid eversion, stabilization, slit-lamp aiming, equivalent spot count) using identical laser settings, but with minimal power (50 mW, duration 10 ms) and beam offset to the adjacent non-vascular periorbital skin, ensuring no energy delivery to eyelid margin vessels, and preserving the device operational sound, laser light, and foot pedal activation. No laser energy was delivered to eyelid margin vasculature in the sham treatment, and no visible tissue reaction or blanching was observed during the procedure. The anesthesia and cleaning procedures were identical.
  Interventions: Device: Sham treatment

INTERVENTIONS:
Procedure: laser light — laser photocoagulation of the telangiectatic vessels of the lower eyelid margin with a slit lamp-based 532 nm optically pumped dual- diode solid-state subthreshold (SP-Mode) laser system
  Arms: Laser Group
Device: Sham treatment — Sham treatment replicated all procedural steps (eyelid eversion, stabilization, slit-lamp aiming, equivalent spot count) using identical laser settings, but with minimal power (50 mW, duration 10 ms) and beam offset to the adjacent non-vascular periorbital skin, ensuring no energy delivery to eyelid margin vessels, and preserving the device operational sound, laser light, and foot pedal activation. No laser energy was delivered to eyelid margin vasculature in the sham treatment, and no visible tissue reaction or blanching was observed during the procedure. The anesthesia and cleaning procedures were identical.
  Arms: Control Group

SUMMARY:
The modern treatment of meibomian gland dysfunction(MGD) is based on anti-inflammatory drops or oral antibiotics for decreasing dry eye disease (DED) associated inflammation, warm compresses for liquefying the thicker meibum, and lid hygiene for reducing the bacterial overload. But, such treatments have shown limited effectiveness to a large proportion of patients with MGD, due to the multifactorial background of the disease. Thus, alternative approaches aiming at different aspects of the DED pathophysiology are needed.

Elimination of posterior lid-margin hyperemia with telangiectasia could be a treatment target for reducing the secretion of inflammatory mediators in the course of MGD. Using the mechanism of photocoagulation via selective thermolysis, laser light could contribute to the destruction of abnormal vessels at the posterior lid-margin and thus, the reduction of inflammation. Recently, sub-threshold (micropulse) laser photocoagulation was introduced in ophthalmology and offers significant clinical advantages compared to conventional continuous wave (CW) approach, preventing laser induced thermal damage and related treatment side effects.

This study investigates the effect of sub-threshold (micropulse) laser treatment for dry eye disease due to meibomian gland dysfunction combined with increased eyelid margin vascularity.

ELIGIBILITY:
Inclusion criteria were:

* chief complaint of at least one of the following symptoms: dryness, foreign-body sensation, burning, and tearing for 3 months
* diagnosis of DED secondary to MGD with eyelid margin telangiectasias in both eyes
* a baseline Ocular Surface Disease Index (OSDI) score ≥ 40
* tear break-up time (TBUT) ≤ 5 seconds
* corneal fluorescein staining ≥ 6 as per the National Eye Institute (NEI) grading scale for corneal staining.

Exclusion criteria were:

* history of ocular trauma or surgery
* use of any treatment for DED or MGD other than artificial tears within the past 3 months
* active allergy, infection, or inflammatory disease at the ocular surface unrelated to DED or MGD
* lacrimal drainage system anomalies
* contact lens wear
* use of any systemic or topical anti-inflammatory medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-07-18 (Actual)

PRIMARY OUTCOMES:
Tear Break Up Time (TBUT) | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  Using a slit-lamp biomicroscope with cobalt blue illumination, the time interval between the last complete blink and first appearance of a dark dry spot on the corneal surface was measured using a digital stopwatch. The test was repeated three times consecutively, and the mean TBUT was recorded

SECONDARY OUTCOMES:
Ocular Surface Disease Index (OSDI) | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  The scoring system ranges from 0 to 100 and categorizes the ocular surface condition into normal (0-12), mild (13-22), moderate (23-32), or severe dry eye (≥ 33).15 OSDI questionnaire was administered once per patient to assess subjective symptom severity at each visit, whereas all other parameters were evaluated separately for each eye.
Lower Eyelid Tear Meniscus Height | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  height (μm) via Anterior Segment Swept-Source Optical Coherence Tomography
Lower Eyelid Tear Meniscus Depth | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  depth (μm) via Anterior Segment Swept-Source Optical Coherence Tomography
Meibomography | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  scale (0,1,2,3). Higher values represent greater disability.
Best Corrected Visual Acuity (BCVA) | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively
  using Snellen charts, which was converted to logMAR values for statistical analysis purposes.
Schirmer test | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  under topical anesthesia standardized Schirmer strips were gently inserted into the lateral third of the lower eyelid margin, and the length of wetting (in millimeters) on the strip was recorded after 5 minutes
Eyelid margin vascularity | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  via slit-lamp biomicroscopy and graded on a 4-point scale as 0 (no visible telangiectasia), 1 (mild telangiectasia with few dilated vessels), 2 (moderate telangiectasia with several visible vessels), and 3 (severe telangiectasia with numerous engorged vessels and marked redness).
corneal staining and the conjunctival injection | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively
  using fluorescein dye, according to the National Eye Institute (NEI) scale
Conjunctivochalasis | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  graded by the number and height of conjunctival folds using a slit lamp as 0 (no persistent folds), 1 (one small fold), 2 (two or more folds not higher than the tear meniscus), and 3 (multiple folds higher than the tear meniscus)
Meibomian gland (MG) expressibility | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively.
  by applying standardized digital pressure to the central third of the lower lid, graded as 1 (light), 2 (moderate), or 3 (heavy pressure required).
secretion quality | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively
  0 (clear), 1 (cloudy), 2 (granular), or 3 (toothpaste-like).

OTHER OUTCOMES:
Posterior margin irregularity, hyperkeratosis, lash loss, anterior blepharitis, tear debris, and tear foam | The subjects were evaluated at five different time points: (a) 1 day preoperatively (baseline), (b) 2 weeks (W2), (c) 4 weeks (W4), (d) 8 weeks (W8), and (e) 12 weeks (W12) postoperatively
  as absent (normal) or present (abnormal).

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Kappos, MD, Principal Investigator — Naval Hospital, Athens
Locations (2):
- Greece (2):
  - Naval Hospital of Athens, Athens
  - First Department of Ophthalmology, National and Kapodistrian University of Athens, Athens, Greece, Athens

IPD SHARING:
Plan to Share IPD: No